CLINICAL TRIAL: NCT04737356
Title: SIA - Internet-administered CBT for Adolescents With Low Self-esteem
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Gerhard Andersson, Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIA
Record Dates: First submitted 2021-01-28; First posted 2021-02-03 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Self Esteem
Keywords: cognitive behavior therapy
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavior Therapy (Experimental): Therapist-Guided Internet based Cognitive Behavior Therapy
  Interventions: Behavioral: Cognitive behavior therapy
- Wait-list control (No Intervention): Wait-list control participants will receive the same treatment at the end of the study period.

INTERVENTIONS:
Behavioral: Cognitive behavior therapy — Internet-based CBT intervention based on CBT theory as well as self-determination therapy for low self-esteem among adolescents.
  Arms: Cognitive Behavior Therapy

SUMMARY:
The study will investigate a novel CBT based treatment approach for low self-esteem among adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Low self-esteem, as indicated by rating of < 20 the Rosenberg Self-Esteem Scale.
* Age between 15 and 19 years old.
* Access to a computer, smartphone, or tablet with internet access.
* Write and speak Swedish.
* In case of use of psychotropical medication, a stable dose for the past three months prior to registration and no planned changes during the treatment.

Exclusion Criteria:

* Other ongoing psychological treatment that affects the treatment received in the study.
* No comorbid severe depressive symptoms and no suicidal plans.
* Ongoing alcohol use disorder, as indicated by Alcohol Use Disorders Identification Test (AUDIT).
* Severe psychiatric comorbidities (e.g. psychosis, anorexia nervosa) that requires specialist care within the regular psychiatric care.

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Change in Rosenberg Self-Esteem Scale | Before treatment, after 3 weeks, after 7 weeks and follow-up at 12 months after treatment termination.
  A 10-item measure of self-esteem. Sum scores range between 0-30. A higher score indicates a higher self-esteem.

SECONDARY OUTCOMES:
Change in Brunnsviken Brief Quality of Life Questionnaire | Before treatment, after 7 weeks and follow-up at 12 months after treatment termination.
  Measure of subjective quality of life. Sum scores can range between 0 and 96. Higher scores indicate a higher quality of life.
Change in Robson Self-concept Questionnaire | Before treatment, after 7 weeks and follow-up at 12 months after treatment termination.
  A 30-item measure of self-esteem. Sum scores range between 0-210. A higher score indicates a higher self-esteem.
Change in Self-Compassion Scale Short Format | Before treatment, after 7 weeks and follow-up at 12 months after treatment termination.
  A 12-item measure of self-compassion. Sum scores range between 1-5. A higher score indicates higher self-compassion.
Change in Performance based self-esteem Scale | Before treatment, after 7 weeks and follow-up at 12 months after treatment termination.
  A 4-item measure of performance based self-esteem. Sum scores range between 4-20. A higher score indicates a higher performance based self-esteem.
Change in Patient Health Questionnaire | Before treatment, after 7 weeks and follow-up at 12 months after treatment termination.
  A 9 item measure of depressive symptoms. Sum scores range from 0-27. A higher score indicates more depressive symptoms.
Change in Generalised Anxiety Disorder 7-item scale | Before treatment, after 7 weeks and follow-up at 12 months after treatment termination.
  Seven item measure of generalized anxiety disorder. Sum score range from 0 to 21, with higher scores indicating more generalized anxiety. Cut-offs for interpretation: 0-5 minimal anxiety, 6-9 mild anxiety, 10-14 moderate anxiety, and 15-21 severe anxiety.
Change in Alcohol Use Disorder Identification Test | Before treatment, after 7 weeks and follow-up at 12 months after treatment termination.
  A 10 item measure of alcohol use disorders. Sum scores range from 0-40. A higher score indicates higher alcohol use.
Change in Rathus assertiveness schedule - 6 | Before treatment, after 7 weeks and follow-up at 12 months after treatment termination.
  Six item measure of assertiveness. Sum score range from -18 to 18. A higher score indicates higher assertiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Andersson, Principal Investigator — Linkoeping University
Locations (1):
- Linköping University, Linköping, Sweden